CLINICAL TRIAL: NCT04156633
Title: Clinical Impact of Rapid Identification of Positive Blood Cultures vs. Internal Laboratory Standard
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01860; qu19Egli2
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Bloodstream Infections
Keywords: MALDI-TOF MS; Biofire FilmArray© Blood Culture Identification (BCID) panel; shotgun metagenomic approach
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- conventional identification methods (controls): Patients with positive blood cultures from 2016 to 2018 receiving a conventional identification methods (controls). The conventional identification method consisted in general of an over-night subculture and subsequent identification of the bacterial pathogen using either biochemical profiling or MALDI-TOF MS.
  Interventions: Diagnostic Test: conventional identification method: biochemical profiling or MALDI-TOF MS
- new identification method (cases)Biofire FilmArray© BCID panel: Patients with positive blood cultures from 2018 and 2019 receiving a new identification method (cases). The new identification method is the Biofire FilmArray© Blood Culture Identification (BCID) panel, a polymerase chain reaction-based method, performed directly from the positive blood culture without the need of subculture to reach single bacterial colonies. The assays allow to identify a panel of 20 most commonly Gram-positive and -negative bacteria and yeast causing blood stream infections. It also allows to determine three resistance genes (mecA, vanA/B and KPC).
  Interventions: Diagnostic Test: new identification method: Biofire FilmArray© BCID panel
- new identification method (cases) WGS approaches: Patients with positive blood cultures from 2018 and 2019 receiving a new identification method (cases). The new identification of positive blood cultures methods in a subset of patients is a whole genome sequencing approach. This so called shotgun metagenomic approach allows to sequence the whole genome (WGS) of pathogens and thereby potentially detect every potential pathogen and also resistance and virulence gene.
  Interventions: Diagnostic Test: new identification method: metagenomic WGS

INTERVENTIONS:
Diagnostic Test: conventional identification method: biochemical profiling or MALDI-TOF MS — Identification of bacteria in positive blood cultures with MALDI-TOF MS from a subculture usually one day after the signal for a positive blood culture appears (from 2016 to 2018)
  Groups: conventional identification methods (controls)
Diagnostic Test: new identification method: Biofire FilmArray© BCID panel — The Biofire FilmArray© BCID Panel is performed directly from the positive blood culture without the need of subculture to reach single bacterial colonies (from 2018 and 2019)
  Groups: new identification method (cases)Biofire FilmArray© BCID panel
Diagnostic Test: new identification method: metagenomic WGS — shotgun metagenomic approach allows to sequence the whole genome (WGS) of pathogens and thereby potentially detect every potential pathogen and also resistance and virulence gene (from 2018 and 2019)
  Groups: new identification method (cases) WGS approaches

SUMMARY:
In this before-after study, different new methods for bacterial species identification from positive blood cultures will be compared towards historic controls. All samples are analyzed within the routine workflow for bacterial species identification and antibiotic resistance profiling. Patients with positive blood cultures from 2016 to 2018 receiving a conventional identification methods (controls) will be compared to patients from 2018 and 2019 with a new identification method (cases). The conventional identification method consisted in general of an over-night subculture and subsequent identification of the bacterial pathogen using either biochemical profiling or Matrix-assisted Laser-Desorption/Ionization Time-of-Flight (MALDI-TOF MS). The new identification of positive blood cultures methods include (i) either the newly introduced Biofire FilmArray© Blood Culture Identification (BCID) panel or (ii) in a subset of patients whole genome sequencing (WGS) approaches.

ELIGIBILITY:
Inclusion Criteria:

* patients with positive blood cultures hospitalized between August 2016 and October 2019
* documented refusal of the general consent

Exclusion Criteria:

* outpatients
* patients hospitalized in other hospitals
* patients with known bacteremia diagnosed in another hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with positive blood cultures hospitalized at the university hospital Basel between August 2016 and October 2019 are included.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Time to optimal antibiotic treatment in hours from positive blood cultures (hours) | 24 hours from collection of blood cultures
  Time from blood draw for blood culture testing to start of optimal antibiotic treatment (hours)

SECONDARY OUTCOMES:
Time to effective antibiotic treatment in hours from positive blood cultures (hours) | 24 hours from collection of blood cultures
  Time from blood draw for blood culture testing to start of effective antibiotic treatment (hours)
all-cause in hospital mortality (number) | from admission to hospital until release from hospital (approximately 30 days)
  all-cause in hospital mortality (number)
duration on ICU in days | from admission to ICU until release from ICU (approximately 20 days)
  duration on ICU in days
time to Gram staining and resistance profile from positive blood cultures (hours) | 24 hours from collection of blood cultures
  time to Gram staining and resistance profile from positive blood cultures (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD Dr. med, Principal Investigator — Division of Clinical Bacteriology & Mycology; University Hospital Basel
Locations (1):
- Division of Clinical Bacteriology & Mycology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Agnetti J, Buchler AC, Osthoff M, Helfenstein F, Weisser M, Siegemund M, Bassetti S, Bingisser R, Schaefer DJ, Clauss M, Hinic V, Tschudin-Sutter S, Battig V, Khanna N, Egli A. Identification of microorganisms by a rapid PCR panel from positive blood cultures leads to faster optimal antimicrobial therapy - a before-after study. BMC Infect Dis. 2023 Oct 26;23(1):730. doi: 10.1186/s12879-023-08732-9. PMID 37884860